CLINICAL TRIAL: NCT01987375
Title: Phase I, Open-label Study Evaluating the Safety and Pharmacokinetics of Escalating Doses of Cetuximab-IRDye800 as an Optical Imaging Agent to Detect Cancer During Surgical Procedures
Brief Title: Cetuximab IRDye800 Study as an Optical Imaging Agent to Detect Cancer During Surgical Procedures
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: logistics
Sponsor: Eben Rosenthal (Other)
Responsible Party: Sponsor-Investigator, Eben Rosenthal, Professor of Otolaryngology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-35068; ENT0049 (Other: OnCore)
Record Dates: First submitted 2013-10-08; First posted 2013-11-19 (Estimated); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Head and Neck Cancer
Keywords: HNSCC; Imaging
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab-IRDye800 Participants (Experimental): Participants who received the study drug cetuximab-IRDye800, following a loading dose of unlabeled cetuximab
  Interventions: Drug: Cetuximab-IRDye800

INTERVENTIONS:
Drug: Cetuximab-IRDye800 — a single dose of the study drug following a single loading dose of unlabeled cetuximab

SUMMARY:
This study is an open label, single institution, Phase 1 dose-escalation study to determine the safety profile of cetuximab-IRDye800 used in subjects with head and neck squamous cell carcinoma (HNSCC) that undergo surgery with curative intent. Participants will be given a dose of an approved head and neck cancer drug (Cetuximab) along with an investigational study drug called Cetuximab-IRDye800. Cetuximab-IRDye800 is a drug that is given prior to surgery that attaches to cancer cells and appears to make them visible to the doctor when he uses a special camera during the operation. The investigators are evaluating whether or not the use of the study drug along with the special camera will better identify the cancer while patients are in the operating room.

DETAILED DESCRIPTION:
This study will be a conventional 3+3 phase I study evaluating three escalating dose levels of intravenous infusion of cetuximab-IRDye800 for patients who tolerate a 100 mg test/loading dose of unlabeled cetuximab as part of the screening process. Two cohorts will be added that do not include a 100 mg unlabeled test/loading dose of cetuximab, but will include a 10 mg test dose prior to enrollment. One cohort of 6 patients will be added that includes a 100 mg unlabeled test/loading dose of cetuximab and a fixed 50 mg dose of cetuximab-IRDye800.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy confirmed diagnosis of squamous cell carcinoma of the head and neck.
2. Patients diagnosed with any T stage, any subsite within the head and neck that are scheduled to undergo surgical resection. Patients with recurrent disease or a new primary will be allowed.
3. Planned standard of care surgery with curative intent for squamous cell carcinoma
4. Age ≥ 19 years
5. Have life expectancy of more than 12 weeks
6. Karnofsky performance status of at least 70% or ECOG/Zubrod level 1
7. Have acceptable hematologic status, coagulation status, kidney function, and liver function including the following clinical results:

   * Hemoglobin ≥ 9gm/dL
   * Platelet count ≥ 100,000/mm3
   * Magnesium, potassium and calcium greater than or equal than the lower limit of normal range per institution normal lab values
   * TSH <10 micro International Units/mL

Exclusion Criteria:

1. Received an investigational drug within 30 days prior to first dose of cetuximab-IRDye800
2. Had within 6 months prior to enrollment: MI, CVA, uncontrolled CHF, significant liver disease, unstable angina
3. Inadequately controlled hypertension with or without current antihypertensive medications
4. History of infusion reactions to cetuximab or other monoclonal antibody therapies.
5. Women who are pregnant or breast feeding
6. Patients who have a grade 2 or greater reaction with the test/loading cetuximab dose.
7. Evidence of QT prolongation on pretreatment ECG (greater than 440 ms in males or greater than 450 ms in females).
8. Lab values that in the opinion of the primary surgeon would prevent surgical resection.
9. Patients receiving Class IA (quinidine, procanamide) or Class III (dofetilide, amiodarone, sotalol) antiarrhythmic agents.
10. Patients with TSH>11

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-11; Primary Completion 2017-04-19 (Actual); Study Completion 2017-04-19 (Actual)

PRIMARY OUTCOMES:
Number of subjects in a cohort experiencing a DLT (gr 2 or greater AE considered at least possibly related to study drug & clinically significant by the PI) after receiving cetuximab conjugated to the optical dye IRDye800CW(cetuximab-IRDye800) | 30 days post intervention

SECONDARY OUTCOMES:
Number of subjects with identifiable cancer as compared to surrounding normal tissue by correlating fluorescence with histological evidence of tumor post receipt of cetuximab conjugated to the optical dye, IRDye800CW (cetuximab-IRDye800) | One year post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eben Rosenthal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States